CLINICAL TRIAL: NCT02199327
Title: Clinical Trial to Compare Topical Interferon Alfa 2b And Mitomycin C in Conjunctival-Corneal Intraepithelial Neoplasia
Brief Title: Topical Interferon Alfa 2b and Mitomycin C in Conjunctival-Corneal Intraepithelial Neoplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); University of Guadalajara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2012-785-094
Record Dates: First submitted 2014-07-08; First posted 2014-07-24 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2016-08

CONDITIONS: Conjunctival Intraepithelial Neoplasia; Corneal Intraepithelial Neoplasia
Keywords: Conjunctival-corneal intraepithelial neoplasia; Mitomycin C; Interferon alfa 2b
MeSH Terms: interventions — Mitomycin; Interferon alpha-2; Introns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitomycin C (Active Comparator): Mitomycin C 0.04% 4 times daily for 7 days and 7 days off until resolution of neoplasia (3-6 cycles).
  Interventions: Drug: Mitomycin C
- Interferon alfa 2b (Active Comparator): Interferon alfa-2b 1 million IU/ml 4 times daily until complete resolution of the tumor
  Interventions: Drug: Interferon Alfa-2b

INTERVENTIONS:
Drug: Mitomycin C — Patients treated with mitomycin will be handled by cycles until resolution of the lesion, which according to previous studies is expected between 3 and 6 cycles (between half months and 3 months).
  Other Names: Mutamycin; Mitomycin
  Arms: Mitomycin C
Drug: Interferon Alfa-2b — Patients managed with interferon will be treated for a period ranging from one month to 12 months according to clinical resolution of the lesion. Both groups will be evaluated by at least one year after the resolution of the lesion to determine the presence of recurrences
  Other Names: Urifron; Intron A
  Arms: Interferon alfa 2b

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy of interferon alfa 2b and topical mitomycin C in patients with diagnosis of conjunctival-corneal intraepithelial neoplasia.

DETAILED DESCRIPTION:
The corneal and conjunctival intraepithelial neoplasia is the most common malignant tumor of the ocular surface. Classic treatment is complete excision with safety margins, however, usually the edges are not sharp and difficult clinical differentiation between healthy areas that are not; to this treatment has joined him carrying out cryotherapy bedding and borders . Despite this treatment the recurrence rate ranges from 9-52 %. Antineoplastic drugs have been used either as adjuvant or primary treatment . Among the drugs used the investigators have mitomycin C (MMC) and interferon alpha 2b (INFα 2b).

Controlled clinical trial , single-blind , randomized . Non-probability sampling of consecutive cases. Patients will be assigned to treatment with MMC or INFα2b Periodic clinical evaluations and photos will be made. Time of resolution, resistance and adverse effects will be determined.

Patients treated with mitomycin will be handled by cycles until resolution of the lesion, which according to previous studies is expected between 3 and 6 cycles (between half months and 3 months).

Patients managed with interferon will be treated for a period ranging from one month to 12 months according to clinical resolution of the lesion. Both groups will be evaluated by at least one year after the resolution of the lesion to determine the presence of recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of corneal and conjunctival intraepithelial neoplasia (CIN) with no history of ocular neoplasia

Exclusion Criteria:

* Patients who did not agree to participate in the study.
* Patients with corneal abrasion
* Patients who have the diagnosis of CIN, but are pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12-16 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Therapeutic effect - 100% resolution- with interferon alfa-2b and mitomycin C in patients diagnosed with primary conjunctival-corneal intraepithelial neoplasia | One month to one year
  Patients treated with mitomycin will be handled by cycles until resolution of the lesion, which according to previous studies is expected between 3 and 6 cycles (between half months and 3 months).
  Patients managed with interferon will be treated for a period ranging from one month to 12 months according to clinical resolution of the lesion. Both groups will be evaluated by at least one year after the resolution of the lesion to determine the presence of recurrences.

SECONDARY OUTCOMES:
Adverse effects with topic therapy | One to two years
  Watch as topical treatment is maintained and at least one years after the resolution of the lesion.

OTHER OUTCOMES:
Recurrence of conjunctival-corneal intraepithelial neoplasia | One year
  Watch at least one year after the resolution of the lesion to detect recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Alvarado Beatriz, M.D., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- IMSS Centro Médico de Occidente, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
we intend to publish the results as a scientific article with all results of participants